CLINICAL TRIAL: NCT04264897
Title: Does Insulin Sensitivity Impact the Potential of Metformin to Slow Aging
Brief Title: Antecedent Metabolic Health and Metformin Aging Study
Acronym: ANTHEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Oklahoma (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10699; R01AG064951 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-03

CONDITIONS: Aging; Insulin Sensitivity; Chronic Disease; Mitochondria; Insulin Resistance
Keywords: Blood Glucose Regulation; 5' adenosine monophosphate-activated protein kinase; Healthspan; Skeletal muscle; Mitochondria
MeSH Terms: conditions — Insulin Resistance; Chronic Disease | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled clinical trial of healthy older male and female subjects 40-75 years of age. Subjects will be randomized into one of two groups (metformin or placebo) for a 12-week intervention. The study is double-blinded on placebo versus metformin. The randomization sequence will be stratified by study center (OUHSC or UWM) and baseline insulin status (HOMA-IR <=2.2 [sensitive] versus >=2.5 [resistant]) and will be created using randomly chosen block sizes of four or six. At each center, there will be four groups: insulin sensitive (IS) placebo, IS metformin, insulin resistant (IR) placebo, and IR metformin.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects assigned to the placebo group will receive visually identical pills (silicified microcrystalline cellulose, Micosolle®, K30 povidone, sodium starch glycolate, and magnesium stearate). Only the study statistician and pharmacist will know the metformin versus placebo assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): The investigators use a "ramp up" dosing protocol in which the amount of metformin (Hunter Pharmacy) will begin at 500 mg/day in week 1, increase to 1000 mg/day in week 2, and then to 1500 mg/day in week 3, as tolerated. At week 3 and for the remaining 9 weeks, the dose will remain at 1500 mg/day, which is a standard clinical dose (1500-2000 mg/day). If a subject has gastrointestinal discomfort with 1500 mg/day the dose, the investigators will lower the dose to 1000 mg/day. The investigators will split the dose with 1/2 given in the a.m. and 1/2 in the p.m. and taken with meals to minimize GI discomfort.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Subjects assigned to the placebo group will receive visually identical pills (silicified microcrystalline cellulose, Micosolle®, K30 povidone, sodium starch glycolate, and magnesium stearate).
  The same dosing schedule will be followed as for metformin. The investigators use a "ramp up" dosing protocol in which the amount of placebo (Hunter Pharmacy) will begin at 500 mg/day in week 1, increase to 1000 mg/day in week 2, and then to 1500 mg/day in week 3, as tolerated. At week 3 and for the remaining 9 weeks, the dose will remain at 1500 mg/day. If a subject has gastrointestinal discomfort with 1500 mg/day the dose, the investigators will lower the dose to 1000 mg/day. The investigators will split the dose with 1/2 given in the a.m. and 1/2 in the p.m. and taken with meals to minimize GI discomfort.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Metformin — Metformin (Hunter Pharmacy) following a "ramp up" dosing protocol with a targeted dose of 1500 mg/day for 12 weeks.
  Other Names: Glucophage, Glucophage extended-release, Fortamet, Glumetza, Riomet
  Arms: Metformin
Drug: Placebo oral tablet — Silicified microcrystalline cellulose, Micosolle®, K30 povidone, sodium starch glycolate, and magnesium stearate
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Aging is the number one risk factor for the majority of chronic diseases. There are no pharmaceutical treatments to slow aging and prolong healthspan. The anti-diabetic drug metformin is considered a likely pharmaceutical candidate to slow aging. In this study, the investigators hypothesize that metformin treatment in subjects free of type 2 diabetes will improve insulin sensitivity and glucoregulation in insulin resistant individuals, but will decrease insulin sensitivity and glucoregulation in insulin sensitive subjects. Further, the investigators hypothesize that long-term metformin treatment will remodel mitochondria in a way that decreases mitochondrial function in subjects that are insulin sensitive, but improves mitochondrial function in subjects that are insulin resistant. The investigators will use a dual-site, 12- week drug intervention trial performed in a double-blind, placebo-controlled manner on 148 subjects recruited from two separate sites (Oklahoma Medical Research Foundation (OMRF) and University of Wisconsin-Madison (UWM)). After consent and initial subject screening for chronic disease, subjects will be stratified to insulin sensitive (IS) or insulin resistant (IR) groups. Over a 12- week intervention, half of each group will take metformin and half will take a placebo. Pre- and post--intervention, subjects will complete a series of procedures to assess insulin sensitivity, glucose regulation, and biomarkers of aging. The same subjects will provide a skeletal muscle biopsy pre-- and post-intervention to assess the change in mitochondrial function and mitochondrial remodeling with and without metformin treatment. By completion of this project, the investigators expect to provide evidence that helps further delineate who may benefit from metformin treatment to slow aging.

DETAILED DESCRIPTION:
Although there is epidemiological support for health benefits of metformin in patient populations, it is not clear if these protective effects extend to those free of disease. Therefore, there is a need to perform human studies determining which subjects free of chronic disease benefit from metformin treatment. Retrospective analysis of a randomized, double-blinded clinical trial in our lab revealed that subjects who were insulin sensitive had no effect or negative effects on insulin sensitivity when taking metformin during an exercise training program. These data suggest that in some subjects, metformin has detrimental metabolic outcomes that could accelerate aging. There are data both in support of and refuting that metformin inhibits mitochondrial complex I action and/or mitochondrial remodeling. The overall objective of this trial is to determine if subjects currently free of disease benefit from metformin treatment. There are two critical questions that remain unanswered in human subjects: 1) does antecedent metabolic health influence responses to metformin, and 2) does long-term treatment with metformin lead to mitochondrial remodeling and changes in function. To better understand the translational potential of a clinically relevant dose of metformin for the prevention of chronic conditions, this proposal aims to determine how antecedent metabolic health affects the response to metformin treatment, and identify the relationship between skeletal muscle mitochondrial remodeling and mitochondrial function with metformin treatment. The hypotheses are that: 1) metformin treatment in subjects free of Type 2 diabetes will improve insulin sensitivity and glucoregulation in insulin resistant individuals, but will decrease insulin sensitivity and glucoregulation in insulin sensitive subjects, and 2) long-term metformin treatment will remodel mitochondria in a way that decreases mitochondrial function in subjects that are insulin sensitive, but improves mitochondrial function in subjects that are insulin resistant. To test these hypotheses, a 12-week randomized, double-blind clinical trial will be performed in subjects 40-75 yrs of age, free of disease, and stratified by insulin sensitivity (insulin sensitive and insulin resistant). Pre- and post-training assessments include the hyperinsulinemic- euglycemic clamp to measure hepatic and peripheral insulin sensitivity, continuous glucose monitoring to determine glucoregulation, and proposed blood-based biomarkers of aging. Further, the use of novel stable isotope labeling with proteomic analysis will determine individual and complex-specific mitochondrial remodeling. This approach will be combined with analysis of protein modification and turnover to comprehensively analyze mitochondrial effects of metformin treatment in skeletal muscle. By completion of this project, it is expected that there will be evidence that helps further delineate who may benefit from metformin treatment to slow aging.

ELIGIBILITY:
Inclusion Criteria:

* 40-75 years of age (inclusive)
* Free of chronic disease
* Comprehension of the protocol as indicated by an ability to respond to questions about the study after reading the consent form.
* Able to use and be contacted by telephone.
* Able to speak, read, and understand English, and complete a questionnaire in English
* Independently mobile

Exclusion Criteria:

* Pregnancy
* Heart disease (history, abnormal ECG, abnormal stress ECG)
* Cerebrovascular disease (history)
* Cancer (history)
* Chronic respiratory disease (history, forced expiratory volume at one second/forced vital capacity [FEV1/FVC] < 70, FEV1 < 80% predicted)
* Chronic liver disease (history, alanine transaminase [ALT] > 52 IU/L)
* Diabetes (history, HbA1C ≥ 6.5, fasting blood glucose≥126 mg/dl, oral glucose tolerance test [OGTT] ≥ 200 mg/dl at 2 hrs)
* Impaired kidney function (eGFR ,45 mL/min)
* B12 lab values outside of normal range (<193 or >982 pg/mL)
* Alzheimer's (history)
* Chronic kidney disease (history, abnormal blood kidney panel including serum creatinine > 1.4)
* Problems with bleeding, on medication that prolongs bleeding time (if subject cannot safely stop prior to biopsy)
* Those on glucose lowering drugs
* Those planning to have imaging that requires intravenous contrast dye (within 6 weeks) or are on any of the following medications since they are contraindicated with the use of metformin: Dofetilide, Lamotrigine, Pegvisomant, Somatropin, Trimethoprim, Trospium, Gatifloxacin, Cephalexin, Cimetidine, Dalfampridine
* Tobacco use
* Allergies to lidocaine or metformin

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Mean change in insulin sensitivity measure | Change from baseline to 12 weeks
  Change in insulin sensitivity as determined by a hyperinsulinemic-euglycemic clamp
Mean change in mitochondrial function of the electron transport system measured by complex I activity | Change from baseline to 12 weeks
  Mitochondrial function of the electron transport system

SECONDARY OUTCOMES:
Mean change in daily average glucose measure | Change from baseline to 12 weeks
  5-day continuous glucose monitoring
Mean change in blood-based biomarker measures of aging | Change from baseline to 12 weeks
  HbA1c, glucose, and insulin

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin F Miller, PhD, Principal Investigator — Oklahoma Medical Research Foundation; Adam Konopka, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Oklahoma Health Sciences Center, Oklahoma Shared Clinical and Translational Resources, Oklahoma City, Oklahoma
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results from the trial will be disseminated through presentations at professional meetings and through peer-reviewed publications. Data and other resources will be shared as required by NIH Resource Sharing policies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified data will be shared following the publication of the primary manuscripts for each specific aim from the trial by the trial investigators.
Access Criteria: Researchers interested in accessing de-identified data will contact the trial principal investigators to complete data use agreements and paper/presentation proposals needed for consideration of the proposed research.

REFERENCES:
- [Derived] Kumari S, Bubak MT, Schoenberg HM, Davidyan A, Elliehausen CJ, Kuhn KG, VanWagoner TM, Karaman R, Scofield RH, Miller BF, Konopka AR. Antecedent Metabolic Health and Metformin (ANTHEM) Aging Study: Rationale and Study Design for a Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2022 Dec 29;77(12):2373-2377. doi: 10.1093/gerona/glab358. PMID 34865016